CLINICAL TRIAL: NCT01019902
Title: Impact of Maternal Iron Status on Neonatal Iron Status and Auditory Brainstem Response in the Newborn
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: RSRB00024804; 2008-01857 (Other Grant/Funding Number: NRI)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Anemia
Keywords: iron; pregnancy; adolescents; auditory brainstem responses; anemia; neonate
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — At delivery a 15 mL maternal blood sample, 20 ml cord blood sample and the placenta are collected.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to determine how maternal Fe status influences placental and neonatal Fe status in pregnant adolescents and to assess the impact of the Fe endowment of birth on functional outcomes as assessed by auditory brainstem responses within 48 h of delivery in neonates born to these adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (ages 11-18 y) and their newborns will be eligible to participate if the adolescent is carrying a singleton pregnancy, does not have any preexisting medical complications (such as HIV-infection, eating disorders, hemoglobinopathies, malabsorption diseases, steroid use, substance abuse history, or taking medications known to influence iron homeostasis).

Exclusion Criteria:

* Individuals with pregnancy induced hypertension or elevated diastolic blood pressure (>110) will not be eligible to participate in the study. In addition, adolescents who have been previously treated for lead exposure, or those that have been identified as having elevated blood lead concentrations during childhood, will be excluded from the study.
* Data from infants that experience perinatal asphyxia, pathologic neonatal hyperbilirubinemia, respiratory disease, antibiotic therapy (aminoglycosides), CNS infection, sepsis, congenital or middle or external ear lesions, craniofacial anomalies, chromosomal disorders, TORCH (toxoplasmosis, other infections, rubella, cytomegalovirus infection and herpes simplex infection) or those that were clinically unstable with the first 48 h post-delivery will be excluded from ABR studies. Infants born to mothers with positive drug abuse screens at delivery will also be excluded from further study (these screens are automatically run among this age group). Infants that are identified with hearing deficits at birth using the OAE screening will be excluded from the ABR measures.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant adolescents in Rochester, NY.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2008-10; Primary Completion 2012-11 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Auditory Brainstem Responses (ABR) in Infant | within 24-48 h of birth

SECONDARY OUTCOMES:
Maternal Fe and micronutrient status (folate, B12, Fe, copper and zinc, hemoglobin, hematocrit,transferrin receptor, hepcidin, erythropoietin, ferritin, erythrocyte zinc protoporphyrin/heme ratios and c-reactive protein) | Delivery
Neonatal Fe and micronutrient status | Delivery
Placental Fe/copper/zinc content and expression of key iron transporters. | Delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly O'Brien, PhD, Principal Investigator — Cornell University; Ronnie Guillet, MD, PhD, Principal Investigator — University of Rochester
Locations (1):
- Highland Hospital, Rochester, New York, United States

REFERENCES:
- [Derived] Barad A, Guillet R, Pressman EK, Katzman PJ, Ganz T, Nemeth E, O'Brien KO. Placental ferroportin protein abundance is associated with neonatal erythropoietic activity and iron status in newborns at high risk for iron deficiency and anemia. Am J Clin Nutr. 2024 Jan;119(1):76-86. doi: 10.1016/j.ajcnut.2023.10.022. Epub 2023 Oct 27. PMID 37890671
- [Derived] Delaney KM, Barad A, Castillo LF, Hasund CM, Guillet R, Pressman EK, Katzman PJ, Ganz T, Nemeth E, O'Brien KO. Placental Erythroferrone and Erythropoietin mRNA Expression is not Associated with Maternal or Neonatal Iron Status in Adolescents Carrying Singletons and Adult Women Carrying Multiples. J Nutr. 2023 Jul;153(7):1950-1958. doi: 10.1016/j.tjnut.2023.05.023. Epub 2023 May 28. PMID 37253412
- [Derived] Delaney KM, Guillet R, Fleming RE, Ru Y, Pressman EK, Vermeylen F, Nemeth E, O'Brien KO. Umbilical Cord Serum Ferritin Concentration is Inversely Associated with Umbilical Cord Hemoglobin in Neonates Born to Adolescents Carrying Singletons and Women Carrying Multiples. J Nutr. 2019 Mar 1;149(3):406-415. doi: 10.1093/jn/nxy286. PMID 30770543
- [Derived] Lumish RA, Young SL, Lee S, Cooper E, Pressman E, Guillet R, O'Brien KO. Gestational iron deficiency is associated with pica behaviors in adolescents. J Nutr. 2014 Oct;144(10):1533-9. doi: 10.3945/jn.114.192070. Epub 2014 Aug 13. PMID 25122650
- [Derived] Lee S, Guillet R, Cooper EM, Westerman M, Orlando M, Pressman E, O'Brien KO. Maternal inflammation at delivery affects assessment of maternal iron status. J Nutr. 2014 Oct;144(10):1524-32. doi: 10.3945/jn.114.191445. Epub 2014 Jul 30. PMID 25080540
- [Derived] Jaacks LM, Young MF, Essley BV, McNanley TJ, Cooper EM, Pressman EK, McIntyre AW, Orlando MS, Abkowitz JL, Guillet R, O'Brien KO. Placental expression of the heme transporter, feline leukemia virus subgroup C receptor, is related to maternal iron status in pregnant adolescents. J Nutr. 2011 Jul;141(7):1267-72. doi: 10.3945/jn.110.135798. Epub 2011 May 18. PMID 21593354